CLINICAL TRIAL: NCT00293826
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Dose Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Subcutaneous AMG 108 in Subjects With Rheumatoid Arthritis.
Brief Title: A Multiple Dose Study to Evaluate Subcutaneous AMG 108 in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20050168
Record Dates: First submitted 2006-02-17; First posted 2006-02-20 (Estimated); Last update posted 2010-03-05 (Estimated); Status verified 2010-03

CONDITIONS: Rheumatoid Arthritis
Keywords: ACR criteria; methotrexate; DMARDs; patient reported outcomes; joint assessment
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — AMG 108

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- 1 (Experimental): 196 subjects
  Interventions: Drug: AMG 108
- 3 (Experimental): 196 subjects
  Interventions: Drug: AMG 108
- 2 (Experimental): 196 subjects
  Interventions: Drug: AMG 108
- 4 (Placebo Comparator): 196 subjects
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 108 — 50mg via SC (subcutaneous) injection every 4 weeks
  Arms: 1
Drug: AMG 108 — 250mg via SC (subcutaneous) injection every 4 weeks
  Arms: 3
Drug: AMG 108 — 125mg via SC (subcutaneous) injection every 4 weeks
  Arms: 2
Drug: Placebo — Placebo via SC (subcutaneous) injection every 4 weeks
  Arms: 4

SUMMARY:
The purpose of this study is to determine if AMG 108 in combination with methotrexate is safe and effective in the treatment of rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with active rheumatoid arthritis as diagnosed by meeting ACR classification criteria for at least 6 months.
* Must be taking MTX consecutively for >/= 12 weeks and at a stable dose of methotrexate at 15-25 mg weekly for at least 4 weeks prior to screening

Exclusion Criteria:

* Receipt of commercial or experimental biologic therapies for the treatment of inflammatory disease
* Presence of serious infection
* Class IV rheumatoid arthritis
* Prior or current history of tuberculosis infection or exposure
* Any other DMARDs other than methotrexate within 6 weeks of screening
* Pregnant or nursing
* Receipt of live vaccines within 3 months
* Felty's syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 813 (Actual)
Dates: Start 2006-03; Primary Completion 2007-11 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
ACR20 response | 24 Weeks

SECONDARY OUTCOMES:
Change in subject reported outcomes | 24 Weeks
ACRn, AUC ACRn, ACR50, ACR70, and DAS28 | 24 Weeks
PK parameters | 24 Weeks
Safety endpoints including AEs, SAEs, SIEs, and change in anti-AMG 108 antibody status | 24 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Cardiel MH, Tak PP, Bensen W, Burch FX, Forejtova S, Badurski JE, Kakkar T, Bevirt T, Ni L, McCroskery E, Jahreis A, Zack DJ. A phase 2 randomized, double-blind study of AMG 108, a fully human monoclonal antibody to IL-1R, in patients with rheumatoid arthritis. Arthritis Res Ther. 2010;12(5):R192. doi: 10.1186/ar3163. Epub 2010 Oct 15. PMID 20950476
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf